CLINICAL TRIAL: NCT02535403
Title: Internet-based Cognitive Behavioral Therapy (CBT) for Adolescents With Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chilled Out DK
Record Dates: First submitted 2015-08-21; First posted 2015-08-28 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

ARMS (2):
- ICBT (Experimental): 14 weeks of internet-based cognitive behavioral therapy with therapist support
  Interventions: Behavioral: ICBT
- Wait-list (No Intervention): 14 weeks wait-list control

INTERVENTIONS:
Behavioral: ICBT
  Arms: ICBT

SUMMARY:
Cognitive behavioral therapy (CBT) is a well-documented and effective method for the treatment of children and adolescents with anxiety disorders. Lately there has been an increase in the development and use of internet-based CBT programs (ICBT), as a means to reduce costs and enhance accessibility of psychological interventions. ICBT has proven efficacious towards adults with anxiety disorders. Research in the field of ICBT with children and adolescents is still in its infancy though and to date, no program targeting anxiety disorders has been developed nor evaluated in Denmark. The primary objective of this study is to investigate the efficacy of a newly developed internet-based treatment program for adolescents with anxiety disorders. The effect will be examined in a randomized controlled trial comparing ICBT to a wait-list control condition.

DETAILED DESCRIPTION:
Within the context of a research and teaching clinic at the Department of Psychology and Behavioral Sciences, Aarhus University, Denmark, 70 adolescents aged 13-17 with a primary anxiety disorder as assessed by the ADIS C/P will be randomly allocated to either a 3 month wait-list control condition or a treatment condition.

The treatment consists of an internet-based self-help program for adolescents with anxiety disorders called 'Chilled Out', based on material from the well-established manualised group-treatment Cool Kids Program: Adolescent version. It consists of 8 CBT-inspired modules of approximately 30 minutes each distributed over a 14-week period. The program is interactive using a combination of different media (text, audio, illustrations, cartoons, and videos) to deliver psychoeducation and CBT-inspired techniques, activities and exercises for adolescents to manage their anxiety. In addition, the adolescent will receive a limited amount of therapist support calls.

Participants (youth and parents) are assessed with semi-structured diagnostic interviews and self-report measures before treatment, after 14 weeks (post treatment) and 3 months after treatment (follow-up).

Participants are assessed at pre, post and 3-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* a primary diagnosis of separation anxiety disorder, generalized anxiety disorder, social phobia, specific phobia, obsessive compulsive disorder or panic disorder
* age between 13 and 17 years
* ability to read and write in Danish
* direct access to a home computer and internet

Exclusion Criteria:

* high degree of comorbid depression (CSR above 5 as measured with ADIS-IV)
* substance abuse
* current self-harm or suicidal ideation
* pervasive developmental disorder
* learning disorder
* intellectual disability
* psychotic symptoms

All participants are asked not to make changes to their medication status during the course of the trial

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in The Anxiety Disorder Interview Schedule for DSM-IV, Parent and Child Versions (ADIS-IV c/p) | Pre- (baseline) and post- (14 weeks) treatment + 3 months follow-up
  Measures clinician rated anxiety symptoms through Clinician Severity Rating (CSR)
Change in Spence Child Anxiety Scale (SCAS-C/P) | Pre- (baseline) and post- (14 weeks) treatment + 3 months follow-up
  Measures self-rated youth anxiety symptoms

SECONDARY OUTCOMES:
Change in Children's Anxiety Life Inference Scale (CALIS) | Pre- (baseline) and post- (14 weeks) treatment + 3 months follow-up
  Measures life interference and impairment associated with the anxiety disorder(s) as assessed by parents and youths
Change in Self-Efficacy Questionnaire for Children (SEQ-c) | Pre- (baseline) and post- (14 weeks) treatment
  Measures youth self-efficacy
Change in the Short version of the Mood and Feelings Questionnaire (S-MFQ-c/p) | Pre- (baseline) and post- (14 weeks) treatment
  Measures youth depressive symptoms as assessed by parents and youths
Change in WHO Quality of Life (5 items) | Pre- (baseline) and post- (14 weeks) treatment + 3 months follow-up
  A short version of The World Health Organization Quality of Life questionnaire (WHOQOL) measuring youth quality of life
Change in Strength and Difficulties Questionnaire for Youth (SDQ) | Pre- (baseline) and post- (14 weeks) treatment
  Measures youth strengths and difficulties as assessed by youths and parents
Change in Working Alliance Inventory - Short form (WAI-S) | Mid- (4 and 8 weeks) and post- (14 weeks) treatment
  Measures the therapeutic alliance between youth and therapist
Experience of Service Questionnaire (ESQ) | Post- (14 weeks) treatment
  Measures youths' and parents' satisfaction with the treatment
Adherence to the program I | Post- (14 weeks) treatment
  Degree of program completion (number of completed modules)
Adherence to the program II | Post- (14 weeks) treatment
  Total amount of log ins to the program
Adherence to the program III | Post- (14 weeks) treatment
  Average time spent per week on program relevant activities (online)
Adherence to the program IV | Post- (14 weeks) treatment
  Average time spent per week on program relevant activities (offline)
Parent support | Post- (14 weeks) treatment
  Parents' average time spent per week helping their child with program relevant activities (on- and offline)

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Aarhus, Denmark

REFERENCES:
- [Derived] Stjerneklar S, Hougaard E, McLellan LF, Thastum M. A randomized controlled trial examining the efficacy of an internet-based cognitive behavioral therapy program for adolescents with anxiety disorders. PLoS One. 2019 Sep 18;14(9):e0222485. doi: 10.1371/journal.pone.0222485. eCollection 2019. PMID 31532802